CLINICAL TRIAL: NCT03846219
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Phase 2 Trial Assessing the Effect of IMU-838 on Disease Activity, as Measured by Magnetic Resonance Imaging (MRI), as Well as Safety and Tolerability in Patients With Relapsing-remitting Multiple Sclerosis (RRMS)
Brief Title: MRI Trial to exPlore the efficAcy and Safety of IMU-838 in Relapsing Remitting Multiple Sclerosis (EMPhASIS)
Acronym: EMPhASIS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunic AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2-IMU-838-MS; 2018-001896-19 (EudraCT Number)
Record Dates: First submitted 2019-01-21; First posted 2019-02-19 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis (RRMS)
Keywords: RRMS; Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: This is a Phase 2 multicenter, double-blind, placebo-controlled, randomized, parallel-group trial to assess the efficacy and safety of 2 once-daily oral doses of IMU-838 (30 mg/day and 45 mg/day) in the main study (10 mg/day for the patients in the substudy) in patients with RRMS and evidence of active disease. The trial consists of a screening period, a blinded 24-week main treatment period, and an optional initially blinded, then open-label extended treatment period of up to 9.5 years.
  The trial includes 2 patient cohorts:
  * Cohort 1 main trial: main Phase 2 trial with assessment of primary and key secondary endpoints.
  * Cohort 2 sub-trial: additional sub-trial with a small double-blind, placebo-controlled, randomized, parallel-group assessment of 10 mg/day IMU-838 dose to provide additional data for pharmacodynamic modelling.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial participants, treating and evaluating physicians, central MRI readers and all other personnel directly involved in the conduct of the trial will be blinded to treatment assignments during the main treatment period and for the initial time of the extended treatment period. The evaluating physician will also be blinded to any clinical outcome or treatment change.
  Once the results of the main treatment period are available, treating physicians, participants, and other involved personnel, except for the evaluating physician, will be unblinded. The evaluating physician will remain blinded to patients' clinical characteristics and treatment assignment during the entire clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IMU-838 (30 mg/day) (Experimental): IMU-838 tablet containing 15 mg Vidofludimus calcium (IM90838). Once-daily oral dose of 30 mg consists of 2 tablets IMU-838.
  Duration: until the end of the main treatment period (24 weeks). In the optional extended treatment period, patients were randomized to receive either 30 mg/day or 45 mg/day IMU-838 (up to 9.5 years for the main trial).
  Interventions: Drug: IMU-838 (30 mg/day)
- IMU-838 (45 mg/day) (Experimental): Tablet containing 22.5 mg Vidofludimus calcium (IM90838). Once-daily oral dose of 45 mg consists of 2 tablets.
  Duration: until the end of the main treatment period (24 weeks). In the optional extended treatment period, patients were randomized to receive either 30 mg/day or 45 mg/day IMU-838.
  Interventions: Drug: IMU-838 (45 mg/day)
- Placebo (Placebo Comparator): Tablet containing no active ingredient. The placebo tablets will be identical to the IMU-838 tablets in terms of appearance, constitution of inactive ingredients, and packaging. Once-daily oral dose consists of 2 active compound-free tablets.
  Duration: until the end of the main treatment period (24 weeks). The placebo is not applicable in the optional extended treatment period, in which participants who were receiving placebo in the main treatment period were re-randomized to IMU-838 for the extended treatment period.
  Interventions: Drug: Placebo
- IMU-838 (10 mg/day) - Cohort 2 (Experimental): Cohort 2 sub-trial: additional sub-trial with a small double-blind, placebo-controlled, randomized, parallel-group assessment of a low IMU-838 dose (i.e. 10 mg/day) to provide additional data for pharmacodynamic modelling.
  Tablet containing 5 mg Vidofludimus calcium (IM90838). Once-daily oral dose of 10 mg consists of 2 tablets.
  Duration: until the end of the main treatment period (24 weeks). In the optional extended treatment period, patients were randomized to receive either 30 mg/day or 45 mg/day IMU-838 (up to 8.5 years for the cohort 2 sub-trial).
  Interventions: Drug: IMU-838 (10 mg/day)

INTERVENTIONS:
Drug: IMU-838 (30 mg/day) — * Main treatment period: All patients will receive half the assigned dose during the first 7 days of the main treatment period (one 15 mg tablet IMU-838 daily) and then start taking the full assigned dose from Day 7 onwards (two 15 mg tablets IMU-838 once daily).
  * Optional extended treatment period (optional): Participants who were re-randomized to a 30 mg/day dose will take the full assigned dose which consists of two 15 mg tablets IMU-838 once daily.
  Other Names: Vidofludimus Calcium, Oral Tablet (30 mg/day)
  Arms: IMU-838 (30 mg/day)
Drug: IMU-838 (45 mg/day) — * Main treatment period: All patients will receive half the assigned dose during the first 7 days of the main treatment period (one 22.5 mg tablet per day) and then start taking the full assigned dose from Day 7 onwards (two 22.5 mg tablets once daily).
  * Optional extended treatment period (optional): Participants who were re-randomized to a 45 mg/day dose will take the full assigned dose of two 22.5 mg tablets IMU-838 once daily.
  Other Names: Vidofludimus Calcium, Oral Tablet (45 mg/day)
  Arms: IMU-838 (45 mg/day)
Drug: Placebo — * Main treatment period (Cohort 1 and Cohort 2): All patients will receive 1 tablet per day during the first 7 days of the main treatment period and then start taking 2 tablets once daily from Day 7 onwards.
  * Optional extended treatment period: Placebo not applicable as participants were re-randomized to a 30 mg/day dose or a 45 mg/day dose.
  Arms: Placebo
Drug: IMU-838 (10 mg/day) — * Main treatment period for Cohort 2: All patients will receive half the assigned dose during the first 7 days of the main treatment period (one 5 mg tablet per day) and then start taking the full assigned dose from Day 7 onwards (two 5 mg tablets once daily).
  * Optional extended treatment period (not applicable to Cohort 2): IMU-838 10 mg/day not applicable.
  Other Names: Vidofludimus Calcium, Oral Tablet (10 mg/day)
  Arms: IMU-838 (10 mg/day) - Cohort 2

SUMMARY:
This is a Phase 2 multicenter, double-blind, placebo-controlled, randomized, parallel-group trial to assess the efficacy and safety of 2 once-daily oral doses of IMU-838 (vidofludimus calcium), a small molecule inhibitor of dihydroorotate dehydrogenase (DHODH), 30 mg/day and 45 mg/day in the main study, cohort 1 (and 10 mg/day for the patients in the cohort 2 substudy), in patients with RRMS and evidence of active disease.

The trial consists of a screening period, a blinded 24-week main treatment period, and an optional initially blinded, then open-label extended treatment period of up to 9.5 years.

About 40 centers are planned to participate in Romania, Bulgaria, Ukraine, and Poland; potential additional centers in Hungary and Croatia were not used. The study started with 195 patients in the main group (cohort 1) planned to be randomized 1:1:1 to treatment with 30 mg/day or 45 mg/day IMU-838, or placebo (65 patients each) in the main treatment period. During the extended treatment period, patients were initially re-randomized so that patients previously on placebo were re-randomized 1:1 to treatment with 30 g/day or 45 mg/day IMU-838, all other patients were re-randomized to the same treatment they previously received.

With approval of Protocol Version 3.0, a sub-study patient group (cohort 2) has been added with up to 60 patients, randomized to placebo or 10 mg IMU-838 for 24 weeks after which the option is available to continue into the extended treatment period and the recommended dose of 30 mg/day. However, based on discussion between investigator and patient 45 mg/day IMU-838/day may also be used.

ELIGIBILITY:
Inclusion criteria for the main treatment period

1. Male or female patient (age ≥18 to 55 years, inclusive)
2. Diagnosis of RRMS according to the revised McDonald criteria (2017) Note: The diagnosis of MS (including "dissemination in time") must have been established before the patient is screened for the trial.
3. Disease activity evidenced

   * by either at least 2 relapses in the last 24 months, or at least 1 relapse in the last 12 months before randomization (relapses must have been assessed and documented by a physician in the patient files), AND
   * ≥1 documented Gd+ MS-related brain lesion, in the last 6 months before informed consent (date of MRI examination as well as copy of MRI report or representative image has to be available and accessible as patient source data at the study site)
4. Expanded Disability Status Scale (EDSS) score between 0 and 4.0 (inclusive) at Screening Visit 1
5. Female patients

   * must be of non-child-bearing potential i.e. surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before Screening Visit 1) or post menopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or
   * if of child-bearing potential, must have a negative pregnancy test at Screening Visit 1 (blood test) and before the first IMP intake (Day 0 urine test). They must agree not to attempt to become pregnant, must not donate ova, and must use a highly effective contraceptive method (see below) together with a barrier method between trial consent and 30 days after the last intake of the of the IMP.

   Highly effective forms of birth control are those with a failure rate less than 1% per year and include:
   * oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraceptives associated with inhibition of ovulation
   * oral, injectable, or implantable progestogen-only hormonal contraceptives associated with inhibition of ovulation
   * intrauterine device or intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * vasectomized partner (i.e. the patient's male partner underwent effective surgical sterilization before the female patient entered the clinical trial and is the sole sexual partner of the female patient during the clinical trial)
   * sexual abstinence (acceptable only if it is the patient's usual form of birth control/lifestyle choice; periodic abstinence [e.g. calendar, ovulation, symptothermal, postovulation methods] and withdrawal are no acceptable methods of contraception)

   Barrier methods of contraception include:
   * Condom
   * Occlusive cap (diaphragm or cervical/vault caps) with spermicidal gel/film/cream/suppository
6. Male patients must agree not to father a child or to donate sperm starting at Screening Visit 1, throughout the clinical trial and for 30 days after the last intake of the IMP. Male patients must also

   * abstain from sexual intercourse with a female partner (acceptable only if it is the patient's usual form of birth control/lifestyle choice), or
   * use adequate barrier contraception during treatment with the IMP and until at least 30 days after the last intake of the IMP, and
   * if they have a female partner of childbearing potential, the partner should use a highly effective contraceptive method as outlined in inclusion criterion 5
   * if they have a pregnant partner, they must use condoms while taking the IMP to avoid exposure of the fetus to the IMP
7. Willingness and ability to comply with the protocol
8. Written informed consent given prior to any trial-related procedure

Inclusion criteria for optional extended treatment period

1. Completed 24 weeks of main treatment
2. Baseline MRI and Week 24 MRI, as well as 2 additional post-dose MRIs

Continuation criteria for optional extended treatment period

1. In case the initial Week 24 MRI was not evaluated at least partially assessable, availability of a repeated Week 24 MRI
2. Week 24 MRI (initial or repeated one, if applicable) evaluated at least partially assessable

Exclusion criteria

MS-related exclusion criteria

1. Any disease other than MS that may better explain the signs and symptoms, including history of complete transverse myelitis
2. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from these
3. Clinical signs or presence of laboratory findings suggestive for neuromyelitis optica (NMO) spectrum disorders or MOG-associated encephalomyelitis (i.e. presence of anti-NMO [aquaporin-4] antibodies or anti-MOG-antibodies)
4. MS types other than RRMS
5. Any MRI finding, atypical for MS, including but not limited to a longitudinally extensive spinal cord lesion
6. Any active and uncontrolled coexisting autoimmune disease, other than MS (except for type 1 diabetes mellitus and inflammatory bowel disease)
7. An MS relapse within 30 days before Screening Visit 1 and/or during the screening period (until Day 0)

   Therapy exclusion criteria
8. Any previous or current use of the following MS treatments: monoclonal antibodies (natalizumab, alemtuzumab, daclizumab, ocrelizumab, anti-CD4, rituximab or belimumab, including their biosimilars), total lymphoid irradiation, bone marrow transplantation, stem cell transplantation, or any use of DHODH inhibitors, including teriflunomide (Aubagio™) or leflunomide (Arava™)
9. Any use of the following MS treatments within 12 months before the date of informed consent: any cytokine (other than interferon) or anti-cytokine therapy, intravenous immunoglobulin, mitoxantrone, cytotoxic or immunosuppressive therapy (including, but not limited to azathioprine and cyclophosphamide, excluding only systemic corticosteroids or adrenocorticotrophic hormone [ACTH]), tofacitinib, methotrexate, mycophenolate mofetil, mycophenolate sodium, fingolimod, any calcineurin inhibitors (e.g. tacrolimus, cyclosporine, or pimecrolimus)
10. Any use of the following MS treatments within 30 days before the date of informed consent: interferon-β, glatiramer acetate, dimethyl fumarate and plasmapheresis
11. Within 30 days before the baseline MRI: Use of systemic corticosteroids (intravenous or oral) or ACTH
12. Use of the following concomitant medications is prohibited at Screening Visit 1 and throughout the duration of the trial:

    * any medication known to significantly increase urinary elimination of uric acid, in particular lesinurad (Zurampic™) as well as uricosuric drugs such as probenecid
    * treatments for any malignancy, in particular irinotecan, paclitaxel, tretinoin, bosutinib, sorafinib, enasidenib, erlotinib, regorafenib, pazopanib and nilotinib
    * any drug significantly restricting water diuresis, in particular vasopressin and vasopressin analogs
    * use of rosuvastatin at daily doses higher than 10 mg
13. Use of any investigational product within 8 weeks or 5 x the respective half-life before the date of informed consent, whichever is longer, and throughout the duration of the trial

    Immune response exclusion criteria
14. Conditions negatively affecting the immune response such as previous organ transplant
15. Clinically significantly low lymphocyte and/or neutrophil count (Common Terminology Criteria for AEs Grade of 2 or higher), i.e.

    * lymphocyte count <800/mm³ (0.8 x 109/L), and/or
    * neutrophil count <1,500/mm³ (1.5 x 109/L)
16. History of chronic systemic infections within 6 months before the date of informed consent, including but not limited to tuberculosis, human immunodeficiency virus (HIV), hepatitis B or C
17. Positive IFNγ release assay for Mycobacterium tuberculosis at Screening Visit 1
18. Positive hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (HBcAb), positive HCV-antibody (HCV-Ab) and/or HIV-antigen-antibody test at Screening Visit 1
19. Any live vaccinations within 30 days before the date of informed consent except for the influenza vaccine Other medical history and concomitant disease exclusion criteria
20. Presence of the following laboratory values at Screening Visit 1:

    * platelet count <100,000/mm³ (<100 109/L)
    * serum creatinine >1.5 x ULN
    * total bilirubin, ALT, or GGT >1.5 x ULN
    * Serum uric acid levels at Screening Visit 1 >1.2 x ULN (for women >6.8 mg/dL, for men >8.4 mg/dL)
    * indirect (unconjugated) bilirubin >1.2 x ULN (i.e. >1.1 mg/dL)
21. Known history of nephrolithiasis or underlying condition with a strong association of nephrolithiasis, including hereditary hyperoxaluria or hereditary hyperuricemia
22. History or clinical diagnosis of gout
23. Renal impairment defined as estimated glomerular filtration rate ≤60 mL/min/1.73m²
24. Known or suspected Gilbert syndrome
25. Diagnosis or suspected liver function impairment which may cause fluctuating liver function tests during this trial, as assessed by the investigator
26. History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (New York Heart Association [NYHA] class 3 or 4) Note: NYHA class 3: Cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. NYHA class 4: Cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
27. Clinically relevant, severe pulmonary diseases, uncontrolled hypertension, or poorly controlled diabetes
28. Concurrent malignancy or prior malignancy within the previous 10 years except for the following: adequately-treated non-melanoma skin cancer and adequately-treated cervical cancer
29. History or presence of any major medical or psychiatric illness (such as severe depression, psychosis, bipolar disorder), history of suicide attempt, or current suicidal ideation that in the opinion of the investigator could create undue risk to the patient or could affect adherence with the trial protocol
30. Epilepsy or seizures not adequately controlled by treatment
31. Any other substantial medical condition that in the opinion of the investigator could create undue risk to the patient or could affect adherence with the trial protocol

    General exclusion criteria
32. Current or past (within 12 months of Screening Visit 1) alcohol or drug abuse
33. Any condition that would prevent the patient from undergoing an MRI scan, including:

    * claustrophobic conditions
    * unable to receive Gd-based MRI-contrast agents due to history of hypersensitivity to Gd based contrast agents, or severe renal insufficiency
    * presence of metallic implants incompatible with brain MRI
34. Legal incapacity, limited legal capacity, or any other condition that makes the patient unable to understand the patient information and informed consent form
35. Pregnant or breastfeeding
36. An employee of an investigator or sponsor or an immediate relative of an investigator
37. Patients institutionalized due to judicial or administrative order

Exclusion criteria for optional extended treatment period

1. Any ongoing, clinically significant (as assessed by the investigator) treatment-emergent (started after intake of IMP) AE or laboratory abnormality (including blood chemistry and urinalysis)
2. Significant treatment or trial non-compliance during the main treatment period (as assessed by the investigator), and/or inability or unwillingness to follow instructions by trial personnel
3. Treatment compliance <70% during the main treatment period
4. Significant protocol deviations during the main treatment period that are assessed by the investigator to negatively affect further patient cooperation in this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Muehler, Study Director — Immunic AG
Locations (38):
- Bulgaria (15):
  - MHAT Pulse AD, Department of Neurology Diseases, Blagoevgrad
  - UMHAT "Dr.Georgi Stranski" EAD Pleven Department of Professional Diseases, Pleven
  - MHAT "Heart and brain" EAD Pleven Department of Neurology Diseases, Pleven
  - UMHAT " Kaspela" EOOD, Department of Neurology Diseases, Plovdiv
  - UMHAT "Kanev Ruse", Department of General and Vascular Neurology, Rousse
  - MHATNP "Sveti Naum" EAD, Neurology Clinic for Movement Disorders, First Department of Neurology Diseases, Sofia
  - MHATNPsy "Sveti Naum" EAD, Intensive Therapy Clinic Of Neurology Diseases, Sofia
  - DCC "Neoclinic" EAD, Cabinet Neurology Diseases, Sofia
  - UMHAT "Alexandrovska" EAD, Clinic of Neurology Diseases, Department of Inherited Degenerative and Immunoinflamatori Diseases at Peripheral Nervous System, Sofia
  - UMHAT "Sveti Ivan Rilski" EAD Sofia Clinic of Neurological Diseases, Sofia
  - UMHAT"Alexandrovska"EAD, Department of Degenerative and Immunoinflamatory Disease of the Central Nervous System, Sofia
  - Central Clinical Base-Medical Institute - Ministry of Interior, Neurology Clinic, Sofia
  - Military Medical Academy - Sofia, Clinic of Neurology Diseases, Sofia
  - Military Medical Academy, Clinic of Functional Diagnostics of Nevous System, Sofia
  - UMHAT " Sveta Marina EAD, First Neurology Clinic, Varna
- Poland (5):
  - Nasz Lekarz Ośrodek Badań Klinicznych, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska Paweł Bochniak, Bydgoszcz
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin
  - BioResearch Group Sp. Z o.o, Nadarzyn
  - Centrum Medyczne NeuroProtect, Warsaw
- Romania (5):
  - S.C. Sana Monitoring Srl, Bucharest
  - Spitalul Universitar Elias Bucharesti, Bucharest
  - S.C. Quantum Medical Center Srl, Bucharest
  - Spitalul Clinic Colentina Bucharest, Neurologie 2, Bucharest
  - Spitalul Clinic Cai Ferate Constanta, Constanța
- Ukraine (13):
  - Chernihiv Regional Hospital, Department of Neurology, Chernihiv
  - Dnipropetrovsk Municipal Hospital #5, Neurological Department of the inflammatory and demyelinating diseases of CNS, Dnipro
  - Ukrainian State Research Institute of Medical and Social Problems of Disability of MOH of Ukraine, Dnipro
  - Regional Clinical Hospital, Department of vascular Neurology, Ivano-Frankivsk
  - Kharkiv Regional Clinical Hospital, Department of Neurology, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology NAMSU, Kharkiv
  - Kyiv City Clinical Hospital #4, Department of Neurology, Kyiv
  - Volyn Regional Clinical Hospital, Department of Neurology, Lutsk
  - Poltava Regional Clinical Hospital n.a. Sklifosovskyi, Department of Neurology, Poltava
  - Regional Clinical Centre of Neurosurgery and Neurology, Department #2, Uzhhorod
  - Vinnytsya Regional Psychoneurology Hospital n.a. Yushchenko, Department of Neurology #3, Vinnytsia
  - City Clinical Hospital #2, Department of Neurology, Zaporizhzhya
  - Zaporizhzhya Regional Clinical Hospital, Department of Neurology #1, Zaporizhzhya

REFERENCES:
- [Derived] Fox RJ, Wiendl H, Wolf C, De Stefano N, Sellner J, Gryb V, Rejdak K, Bozhinov PS, Vitt D, Kohlhof H, Slizgi J, Ondrus M, Sciacca V, Muehler AR; EMPhASIS investigators. Safety and Dose-Response of Vidofludimus Calcium in Relapsing Multiple Sclerosis: Extended Results of a Placebo-Controlled Phase 2 Trial. Neurol Neuroimmunol Neuroinflamm. 2024 May;11(3):e200208. doi: 10.1212/NXI.0000000000200208. Epub 2024 Apr 25. PMID 38662979
- [Derived] Fox RJ, Wiendl H, Wolf C, De Stefano N, Sellner J, Gryb V, Rejdak K, Bozhinov PS, Tomakh N, Skrypchenko I, Muehler AR. A double-blind, randomized, placebo-controlled phase 2 trial evaluating the selective dihydroorotate dehydrogenase inhibitor vidofludimus calcium in relapsing-remitting multiple sclerosis. Ann Clin Transl Neurol. 2022 Jul;9(7):977-987. doi: 10.1002/acn3.51574. Epub 2022 Jun 14. PMID 35698927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial consists of a main trial (Cohort 1) and a sub-trial (Cohort 2): Cohort 1 compares 30 mg IMU-838, 45 mg IMU-838 and placebo and assesses the primary and key secondary endpoints; Cohort 2 compares 10 mg/day IMU-838 with placebo. The main trial consists of a blinded 24-week main treatment period and an optional initially blinded, then open-label extended treatment period of up to 9.5 years (currently ongoing).
  Results of the Cohort 1 main treatment period are reported.
Pre-assignment Details: Patients were randomized in a 1:1:1 ratio to once-daily oral treatment with 30 mg IMU-838, 45 mg IMU-838, or matching placebo for 24 weeks. At Week 24 (end-of-main treatment period), patients had the option to continue into the extended treatment period if they met respective eligibility criteria including an magnetic resonance imaging (MRI) scan.
Groups:
- IMU-838 (30 mg/Day): During the main treatment period (24 weeks), patients received once-daily oral doses of 30 mg IMU-838 (2 tablets of 15 mg vidofludimus calcium, IM90838) with an initiation dosing scheme of half the dose (1 tablet per day) during the first 7 days.
- IMU-838 (45 mg/Day): During the main treatment period (24 weeks), patients received once-daily oral doses of 45 mg IMU-838 consisting of 2 tablets of 22.5 mg vidofludimus calcium, IM90838) with an initiation dosing scheme of half the dose (1 tablet per day) during the first 7 days.
- Placebo: During the main treatment period (24 weeks), patients received once-daily oral doses of 2 tablets of placebo with an initiation dosing scheme of half the dose (1 tablet per day) during the first 7 days.
Period: Overall Study
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Started (Patients randomized) | 72 | 69 | 69
Patients Treated | 71 | 69 | 69
Completed | 69 | 65 | 64
Not Completed | 3 | 4 | 5
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Fulfilled hepatoxicity-related stopping rules | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients randomized
Groups:
- IMU-838 (30 mg/Day): During the main treatment period (24 weeks), patients received once-daily oral doses of 30 mg IMU-838 (consisting of 2 tablets of 15 mg vidofludimus calcium [IM90838]).
  All patients received half the assigned dose during the first 7 days of the main treatment period (1 tablet per day) and then started taking the full assigned dose from Day 7 onwards (2 tablets once daily).
- IMU-838 (45 mg/Day): During the main treatment period (24 weeks), patients received once-daily oral doses of 45 mg IMU-838 consisting of 2 tablets of 22.5 mg vidofludimus calcium [IM90838]).
  All patients received half the assigned dose during the first 7 days of the main treatment period (1 tablet per day) and then started taking the full assigned dose from Day 7 onwards (2 tablets once daily).
- Placebo: During the main treatment period (24 weeks), patients received once-daily oral doses of 2 tablets of placebo.
  All patients received 1 tablet per day during the first 7 days of the main treatment period and then started taking 2 tablets once daily from Day 7 onwards.
- Total: Total of all reporting groups
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo | Total
Number analyzed (Participants) | 72 | 69 | 69 | 210
Age, Continuous [Median (Full Range); unit: years] — Population: Full analysis set (FAS, the FAS consisted of all randomized patients who received at least 1 dose of the investigational medicinal product).
  years
    number analyzed (Participants) | 71 | 69 | 69 | 209
    (all) | 38.0 [18 to 55] | 36.0 [21 to 51] | 37.0 [21 to 55] | 36.0 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    number analyzed (Participants) | 71 | 69 | 69 | 209
    Female | 40 | 50 | 46 | 136
    Male | 31 | 19 | 23 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    number analyzed (Participants) | 71 | 69 | 69 | 209
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 71 | 69 | 69 | 209
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    number analyzed (Participants) | 71 | 69 | 69 | 209
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 71 | 69 | 69 | 209
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Patients randomized
  participants
    Romania | 3 | 2 | 1 | 6
    Ukraine | 40 | 36 | 42 | 118
    Poland | 11 | 6 | 9 | 26
    Bulgaria | 18 | 25 | 17 | 60
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Full analysis set
  kg/m^2
    number analyzed (Participants) | 71 | 69 | 69 | 209
    (all) | 23.491 (5.311) | 24.786 (5.067) | 24.462 (4.758) | 24.239 (5.059)
Expanded Disability Status Scale [Mean (Standard Deviation); unit: units on a scale] — The Expanded Disability Status Scale composite rating system ranges from 0 (normal neurological status) to 10 (death due to MS) in 0.5-unit increments. EDSS steps 1.0 to 4.5 refer to a functional status of patients with MS with some limitations within at least one functional system, but still able to walk without any aid. EDSS steps 5.0 to 9.5 are defined by the impairment to walk. Population: Full analysis set
  units on a scale
    number analyzed (Participants) | 71 | 69 | 69 | 209
    (all) | 2.65 (0.83) | 2.56 (0.96) | 2.73 (0.90) | 2.65 (0.90)
Gadolinium enhancing (Gd+) lesions [Mean (Standard Deviation); unit: lesions] — Population: Full analysis set
  lesions
    number analyzed (Participants) | 71 | 69 | 69 | 209
    (all) | 1.4 (2.4) | 0.9 (1.3) | 1.2 (2.1) | 1.2 (2.0)
T2 lesion load [Mean (Standard Deviation); unit: cm^3] — The T2 lesion load per participant was documented in the Case Report Form. In the analysis, a mean across all participants in each arm was calculated. Population: Full analysis set
  cm^3
    number analyzed (Participants) | 71 | 69 | 69 | 209
    (all) | 13.341 (15.079) | 13.918 (12.946) | 11.980 (10.417) | 13.082 (12.940)
MRI field strength [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    number analyzed (Participants) | 71 | 69 | 69 | 209
    1.5 Tesla | 65 | 66 | 67 | 198
    3.0 Tesla | 6 | 3 | 2 | 11
Duration of disease [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    number analyzed (Participants) | 71 | 69 | 69 | 209
    <=4 years | 37 | 37 | 37 | 111
    >4 years | 34 | 32 | 32 | 98

OUTCOME MEASURES:

1. Primary Outcome: Difference Between 45 mg/Day IMU-838 and Placebo in the Cumulative Number of Combined Unique Active (CUA) MRI Lesions
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for baseline volume of T2 lesions, MRI field strength (1.5 or 3.0 Tesla), and baseline number of gadolinium enhancing (Gd+) lesions (0, ≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function. Log transformation of time from first IMP dose to date of last MRI assessment was used as offset term. Mainly due to the differing number of patients with 3.0 Tesla MRI examinations in each treatment arm, the statistical adjustments (to ensure comparabiltiy) for each individual comparison differed and hence the adjusted mean cumulative number of CUA MRI lesions in each arm (e.g. placebo) differed depending on the comparison (45 mg IMU-838 vs placebo, 30 mg IMU-838 vs placebo, or 45 mg vs 30 mg IMU-838).
Time Frame: Up to Week 24
Population: FAS consisting of all randomized patients who received at least 1 dose of the investigational medicinal product (IMP).
Measure: Mean (95% Confidence Interval); unit: CUA MRI lesions
Arm/Group | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 69
CUA MRI lesions | 2.4 [1.1 to 4.9] | 6.3 [2.8 to 13.9]
Statistical Analysis 1: Comparison: IMU-838 (45 mg/Day) vs Placebo; H0: cumulative number of CUA MRI lesions up to Week 24 with 45 mg IMU-838 equal to or higher than that with placebo. A generalized linear model with a negative binomial distribution and logarithmic link function was used. Log transformation of time from 1st IMP dose to date of last MRI assessment was used as offset term. 51 patients per group were necessary to have 80% power to detect a difference of 3.5 in mean event rate with a significance level 0.1, 1-sided; Test type: Superiority; p = 0.0002, generalized linear model — A one-sided alpha level of 0.1 was used; Estimates were adjusted for baseline volume of T2 lesions, MRI field strength (1.5 or 3.0 Tesla), and baseline number of Gd+ lesions (0, ≥1); rate ratio = 0.38, 95% CI 2-sided [0.22 to 0.64] — Rate ratio of 45 mg IMU-838 / placebo

2. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo in the Cumulative Number of Combined Unique Active (CUA) MRI Lesions
Description: This was the key secondary endpoint (hierarchical testing to primary efficacy). MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for baseline volume of T2 lesions, MRI field strength (1.5 or 3.0 Tesla), and baseline number of Gd+ lesions (0, ≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function. Log transformation of time from first IMP dose to date of last MRI assessment was used as offset term. Mainly due to the differing number of patients with 3.0 Tesla MRI examinations in each treatment arm, the statistical adjustments (to ensure comparabiltiy) for each individual comparison differed and hence the adjusted mean cumulative number of CUA MRI lesions in each arm (e.g. placebo) differed depending on the comparison (45 mg IMU-838 vs placebo, 30 mg IMU-838 vs placebo, or 45 mg vs 30 mg IMU-838).
Time Frame: Up to Week 24
Population: FAS consisting of all randomized patients who received at least 1 dose of the IMP.
Measure: Mean (95% Confidence Interval); unit: CUA MRI lesions
Arm/Group | IMU-838 (30 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69
CUA MRI lesions | 4.0 [2.2 to 7.2] | 13.2 [6.6 to 26.4]
Statistical Analysis 1: Comparison: IMU-838 (30 mg/Day) vs Placebo; A generalized linear model with a negative binomial distribution and logarithmic link function was used. Log transformation of time from 1st IMP dose to date of last MRI assessment was used as offset term; Test type: Superiority; p < .0001, Generalized linear model — A hierarchical testing procedure with a one-sided alpha level of 0.1 was used; [statistical method as in outcome 1, analysis 1]; Rate ratio = 0.30, 95% CI 2-sided [0.17 to 0.53] — Rate ratio of 30 mg IMU-838 / placebo

3. Secondary Outcome: Difference Between 45 mg/Day IMU-838 and 30 mg/Day IMU-838 in the Cumulative Number of Combined Unique Active (CUA) MRI Lesions
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for baseline volume of T2 lesions, MRI field strength (1.5 or 3.0 Tesla), and baseline number of Gd+ lesions (0, ≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function. Log transformation of time from first IMP dose to date of last MRI assessment was used as offset term. Mainly due to the differing number of patients with 3.0 Tesla MRI examinations in each treatment arm, the statistical adjustments (to ensure comparabiltiy) for each individual comparison differed and hence the adjusted mean cumulative number of CUA MRI lesions in each arm (e.g. placebo) differed depending on the comparison (45 mg IMU-838 vs placebo, 30 mg IMU-838 vs placebo, or 45 mg vs 30 mg IMU-838).
Time Frame: At Week 24
Population: FAS consisting of all randomized patients who received at least 1 dose of the investigational medicinal product.
Measure: Mean (95% Confidence Interval); unit: CUA MRI lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day)
Number analyzed (Participants) | 71 | 69
CUA MRI lesions | 4.2 [2.5 to 7.1] | 4.4 [2.4 to 8.1]

4. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Mean Number of CUA Lesions Per Patient Per Scan at Weeks 6, 12, 18 and 24
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for MRI field strength (1.5 or 3.0 Tesla) and baseline number of Gd+ lesions (0,≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: CUA MRI lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
CUA MRI lesions
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 1.1 [0.5 to 2.1] | 0.8 [0.4 to 1.8] | 3.2 [1.5 to 6.6]
  Week 12: number analyzed (Participants) | 68 | 65 | 68
  Week 12 | 1.3 [0.7 to 2.3] | 1.2 [0.6 to 2.6] | 3.4 [1.7 to 7.0]
  Week 18: number analyzed (Participants) | 70 | 64 | 65
  Week 18 | 1.3 [0.7 to 2.5] | 0.8 [0.3 to 1.7] | 3.2 [1.5 to 6.6]
  Week 24: number analyzed (Participants) | 69 | 65 | 64
  Week 24 | 1.6 [0.8 to 3.5] | 1.6 [0.6 to 4.4] | 3.7 [1.5 to 9.3]

5. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Cumulative Number of CUA MRI Lesions up to Weeks 6, 12, and 18
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for baseline volume of T2 lesions, MRI field strength (1.5 or 3.0 Tesla), and baseline number of Gd+ lesions (0, ≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function. Log transformation of time from first IMP dose to date of last MRI assessment was used as offset term.
Time Frame: Throughout the main treatment period (Day 0 - Week 18)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: CUA MRI lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
CUA MRI lesions
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 0.8 [0.4 to 1.7] | 0.6 [0.3 to 1.4] | 2.5 [1.1 to 5.5]
  Week 12 | 1.7 [1.0 to 3.0] | 1.6 [0.9 to 3.2] | 5.3 [2.8 to 10.0]
  Week 18 | 2.7 [1.6 to 4.5] | 2.5 [1.4 to 4.6] | 8.0 [4.5 to 14.4]

6. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Volume Changes of T2 Lesions at Weeks 6, 12, 18 and 24 Compared to Baseline
Description: The endpoint was removed in the statistical analysis plan [SAP], since the content was considered the same as the endpoint "T2-lesion load at Weeks 6, 12, 18 and 24 compared to Baseline".
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: This measure was not analyzed because it was determined to be redundant with Outcome Measure 7. No data are available to be reported.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the T2-lesion Load at Weeks 6, 12, 18 and 24 Compared to Baseline
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The percentage change from Baseline in T2 lesion load was calculated.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: % change from Baseline
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
% change from Baseline
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 2.2 [-0.4 to 3.0] | 1.7 [0.3 to 3.6] | 2.4 [0.9 to 4.5]
  Week 12: number analyzed (Participants) | 68 | 65 | 68
  Week 12 | 3.3 [2.2 to 4.9] | 3.4 [2.2 to 5.1] | 4.7 [1.8 to 6.6]
  Week 18: number analyzed (Participants) | 70 | 64 | 65
  Week 18 | 4.9 [2.3 to 7.3] | 4.6 [3.4 to 6.2] | 7.1 [4.8 to 8.9]
  Week 24: number analyzed (Participants) | 69 | 65 | 64
  Week 24 | 6.6 [3.5 to 9.7] | 7.3 [4.2 to 8.7] | 9.0 [7.1 to 12.0]

8. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the T1-lesion Load at Weeks 6, 12, 18 and 24 Compared to Baseline
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The percentage change from Baseline in T1 lesion load was calculated.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: % change from Baseline
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
% change from Baseline
  Week 6: number analyzed (Participants) | 68 | 67 | 63
  Week 6 | -2.9 [-4.9 to -0.9] | -0.4 [-3.3 to 0.8] | -4.2 [-5.7 to -1.2]
  Week 12: number analyzed (Participants) | 67 | 65 | 65
  Week 12 | -4.0 [-5.7 to -1.4] | -1.6 [-4.1 to 0.0] | 0.0 [-2.0 to 0.8]
  Week 18: number analyzed (Participants) | 69 | 64 | 62
  Week 18 | -3.8 [-5.6 to -1.4] | -1.4 [-3.8 to 1.8] | -0.7 [-2.1 to 1.0]
  Week 24: number analyzed (Participants) | 68 | 65 | 61
  Week 24 | -5.7 [-7.6 to -1.7] | -0.9 [-3.6 to 0.0] | -0.8 [-2.3 to 0.7]

9. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Cumulative Number of New Gd+ Lesions up to Weeks 6, 12, 18 and 24
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. Estimates were adjusted for MRI field strength (1.5 or 3.0 Tesla) and baseline number of Gd+ lesions (0, ≥1) using a generalized linear model with a negative binomial distribution and a logarithmic link function. Log transformation of time from first IMP dose to date of last MRI assessment was used as offset term.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: Gd+ lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Gd+ lesions
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 1.0 [0.5 to 2.0] | 0.8 [0.3 to 1.7] | 2.8 [1.3 to 6.2]
  Week 12 | 2.1 [1.2 to 3.7] | 1.7 [0.9 to 3.3] | 6.2 [3.2 to 11.9]
  Week 18 | 3.1 [1.8 to 5.2] | 2.4 [1.3 to 4.5] | 9.1 [4.9 to 16.8]
  Week 24 | 4.5 [2.7 to 7.7] | 4.0 [2.1 to 7.8] | 13.0 [6.8 to 24.5]

10. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Cumulative Number of New T2 Lesions up to Weeks 6, 12, 18 and 24
Description: as for outcome 9
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: T2 lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
T2 lesions
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 0.8 [0.4 to 1.7] | 0.7 [0.3 to 1.5] | 2.6 [1.2 to 5.8]
  Week 12 | 1.8 [1.1 to 3.1] | 1.8 [1.0 to 3.5] | 6.0 [3.2 to 11.2]
  Week 18 | 2.8 [1.7 to 4.5] | 2.7 [1.5 to 4.9] | 8.8 [5.0 to 15.5]
  Week 24 | 4.1 [2.5 to 6.6] | 4.2 [2.3 to 7.7] | 11.9 [6.7 to 21.1]

11. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Cumulative Number of New T1 Lesions up to Weeks 6, 12, 18 and 24
Description: as for outcome 9
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: T1 lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
T1 lesions
  Week 6: number analyzed (Participants) | 69 | 67 | 66
  Week 6 | 0.3 [0.1 to 0.8] | 0.2 [0.1 to 0.6] | 1.1 [0.4 to 3.4]
  Week 12 | 0.6 [0.3 to 1.2] | 0.6 [0.3 to 1.3] | 2.5 [1.1 to 5.6]
  Week 18 | 1.0 [0.6 to 1.9] | 1.0 [0.5 to 1.9] | 3.9 [2.0 to 7.4]
  Week 24 | 1.4 [0.8 to 2.4] | 1.5 [0.8 to 2.9] | 4.7 [2.5 to 8.8]

12. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Number of Patients Without New Gd+ Lesions Over 24 Weeks
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The number of patients who did not develop new Gd+ lesions over the 24-week main treatment period was assessed.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 42 | 34 | 26

13. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Number of Patients Without New or Enlarging T2-weighted Lesions Over 24 Weeks
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The number of patients who did not develop new or enlarging T2 lesions over the 24-week main treatment period was assessed.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 36 | 29 | 22

14. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Number of Patients With CUA Lesions at Week 24
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The number of patients with CUA lesions at Week 24 was assessed.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Patients with observations at Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 65 | 64
Participants | 15 | 19 | 25

15. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Number of Patients With Gd+ Lesions at Week 24
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The number of patients with Gd+ lesions at Week 24 was assessed.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Patients with observations at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 65 | 64
Participants | 10 | 16 | 25

16. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for the Number of Patients With T2 Lesions at Week 24
Description: MRI scans were assessed centrally and adhered to a standardized MRI protocol. The number of patients with T2 lesions at Week 24 was assessed.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Patients with observations in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 65 | 64
Participants | 15 | 18 | 21

17. Secondary Outcome: Differences Between Individual Treatments and Between the Pooled 30 mg/Day and 45 mg/Day Groups and Placebo in the Relapse-related Clinical Endpoints: Mean Annualized Relapse Rate (During Main and Extended Treatment Period)
Description: The adjusted mean annualized relapse rate during the main treatment period was calculated. Estimates were adjusted for baseline number of Gd+ lesions (0, ≥1) using a Poisson model with a logarithmic link function. Log transformation of real exposure time of main treatment period was used as offset term.
  All of the following criteria had to be met for a clinical event to qualify as a relapse:
  1. Neurological deficit, either newly appearing or re-appearing, with abnormality specified by both neurological abnormality separated by at least 30 days from onset of a preceding relapse AND neurological abnormality lasting for at least 24 hours
  2. Absence of fever or known infection (i.e. temperature [axillary, oral, or intra-auricular]
     ≤37.5ºC)
  3. Neurological impairment, defined as either increase in at least one of the functional systems of the EDSS OR increase of the total EDSS score. In both cases, the increase in EDSS had to correlate with the patient's reported symptoms.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Mean (95% Confidence Interval); unit: relapses per person-years
Groups:
- Placebo (Compared With 30 and 45 mg IMU-838); Placebo (Compared With IMU-838 Combined): During the main treatment period (24 weeks), patients received once-daily oral doses of 2 tablets of placebo with an initiation dosing scheme of half the dose (1 tablet per day) during the first 7 days.
- IMU-838 Combined: Groups 30 mg IMU-838 and 45 mg IMU-838 combined
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo (Compared With 30 and 45 mg IMU-838) | IMU-838 Combined | Placebo (Compared With IMU-838 Combined)
Number analyzed (Participants) | 71 | 69 | 69 | 140 | 69
relapses per person-years | 0.39 [0.22 to 0.69] | 0.48 [0.28 to 0.82] | 0.53 [0.32 to 0.89] | 0.43 [0.29 to 0.62] | 0.54 [0.34 to 0.86]

18. Secondary Outcome: Differences Between Individual Treatments and Between the Pooled 30 mg/Day and 45 mg/Day Groups and Placebo in the Relapse-related Clinical Endpoints: Proportion of Relapse-free Patients up to Week 24 and at Extended Periods Thereafter
Description: The proportion of relapse-free patients up to Week 24 was assessed. Patients with no documented relapse and last assessment of relapse before Week 18 were not included. Patients with no documented relapse up to Week 18 and a missing assessment at Week 24 were regarded as relapse-free patients.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Patients analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo | IMU-838 Combined
Number analyzed (Participants) | 70 | 67 | 67 | 137
Participants | 60 | 54 | 51 | 114

19. Secondary Outcome: Differences Between Individual Treatments and Between the Pooled 30 mg/Day and 45 mg/Day Groups and Placebo in the Relapse-related Clinical Endpoints: Time to Relapse at Time of Final Analysis of Main Part
Description: Since only a total of 39 of 209 patients had a relapse up to Week 24, the median time to relapse could not be calculated.
Time Frame: Throughout the main treatment period (Day 0 - Week 24)
Population: Full analysis set
Measure: Median (Full Range); unit: days
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
days | NA [NA to NA] — The median time to relapse could not be calculated. | NA [NA to NA] — The median time to relapse could not be calculated. | NA [NA to NA] — The median time to relapse could not be calculated.

20. Secondary Outcome: Differences Between Treatments in Changes of Disease Activity as Measured by the Mean Change in the Expanded Disability Status Scale (EDSS) as Compared to Baseline During the Main and Extended Period (Every 12 Weeks Starting at Week 12)
Description: The EDSS is a widely used and validated instrument evaluating the functional systems of the CNS to describe disease progression and the efficacy of MS therapy. The composite rating system ranges from 0 (normal neurological status) to 10 (death due to MS) in 0.5-unit increments. An increase in score indicates a worsening.
Time Frame: Baseline, Week 12, and Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
score on a scale
  Week 12: number analyzed (Participants) | 70 | 67 | 69
  Week 12 | -0.01 (0.28) | 0.00 (0.42) | 0.03 (0.38)
  Week 24: number analyzed (Participants) | 67 | 65 | 64
  Week 24 | 0.01 (0.25) | 0.00 (0.39) | 0.08 (0.39)

21. Secondary Outcome: Differences Between Treatments in Changes of Disease Activity as Measured by the Number of Patients With EDSS Progression During the Main and Extended Period (Every 12 Weeks Starting at Week 12, and Cumulatively)
Description: The EDSS is a widely used and validated instrument evaluating the functional systems of the CNS to describe disease progression and the efficacy of MS therapy. The composite rating system ranges from 0 (normal neurological status) to 10 (death due to MS) in 0.5-unit increments. EDSS progression was defined as an increase of the EDSS score compared to Baseline of at least 1.0 point for patients with a baseline EDSS score of 1 to 4.0 or of at least 1.5 points for patients with a baseline EDSS score of 0.
Time Frame: Week 12 and Week 24
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants
  Up to Week 12: number analyzed (Participants) | 70 | 67 | 69
  Up to Week 12 | 6 | 7 | 9
  Up to Week 24: number analyzed (Participants) | 68 | 66 | 65
  Up to Week 24 | 8 | 8 | 15

22. Secondary Outcome: Correlation of MRI-based Assessments With Quartiles of IMU-838 Trough Levels
Description: The cumulative number of CUA MRI lesions up to Week 24 was correlated with quartiles of IMU-838 trough levels at Week 24 of treatment groups IMU-838 30 mg and IMU-838 45 mg.
Time Frame: At Week 24
Population: Patients with observations.
Measure: Mean (Standard Deviation); unit: CUA MRI lesions
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day)
Number analyzed (Participants) | 67 | 64
CUA MRI lesions
  1st quartile of IMU-838 trough level | 1.1 (2.0) | 1.6 (3.1)
  2nd quartile of IMU-838 trough level | 2.2 (4.9) | 1.8 (2.8)
  3rd quartile of IMU-838 trough level | 4.4 (5.8) | 2.0 (2.2)
  4th quartile of IMU-838 trough level | 6.8 (14.7) | 5.3 (9.8)

23. Secondary Outcome: Number of Participants With AEs
Description: The number of patients experiencing treatment-emergent adverse events during the main treatment period was assessed.
Time Frame: Up to 24 weeks
Population: Safety analysis set consisting of all randomized patients who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 32 | 28 | 30

24. Secondary Outcome: Number of Participants With Serious AEs
Description: The number of patients experiencing serious adverse events during the main treatment period was assessed.
Time Frame: Up to 24 weeks
Population: Safety data set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 2 | 0 | 1

25. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities (as Assessed by the Investigator)
Description: Abnormal results in laboratory assessments were assessed by the investigator and classified as clinically significant (yes/no). Clinically significantly abnormal values had to be reported as AE, if not already clinically significantly abnormal at Baseline. Treatment-emergent adverse events related to hematological abnormalities and clinical chemistry abnormalities are reported.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants
  Anemia | 0 | 0 | 1
  Iron deficiency anemia | 0 | 0 | 2
  Leukopenia | 0 | 0 | 1
  Neutropenia | 0 | 0 | 1
  Alanine aminotransferase increased | 1 | 0 | 2
  Aspartate aminotransferase increased | 1 | 0 | 1
  Blood bilirubin increased | 1 | 0 | 0
  Blood creatine phosphokinase increased | 2 | 0 | 0
  Blood creatinine increased | 1 | 0 | 0
  C-reactive protein increased | 0 | 1 | 0
  Hepatic enzyme increased | 1 | 2 | 1
  Lipase increased | 0 | 0 | 1
  Transaminases increased | 0 | 1 | 0
  Hypertriglyceridemia | 1 | 0 | 1

26. Secondary Outcome: Number of Participants With AEs of Special Interest: Red Blood Cell Urine Positive, at Least of Moderate Intensity
Description: The number of patients diagnosed with red blood cell (RBC) urine positive of at least moderate intensity during the main treatment period were assessed.
  The evaluation of RBC in urine was to be solely based on findings from microscopic examinations of urinary sediment and not from dipstick reading only. Therefore, all conspicuous dipstick readings were to be followed up by a microscopic examination of urinary sediment. All findings of RBC in urine per high-powered field (HPF) were to be listed as urinalysis abnormalities but not as an AE, if assessed by the investigator as not clinically significant. The investigator was also to assess any increased RBC in urine as not clinically significant, if there were more likely alternatives to explain this finding.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With AEs of Special Interest: Hematuria
Description: The number of patients diagnosed with hematuria during the main treatment period were assessed.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 0 | 0 | 1

28. Secondary Outcome: Number of Participants With AEs of Special Interest: Retroperitoneal Colicky Pain With Suspected or Confirmed Nephrolithiasis
Description: The number of patients diagnosed with retroperitoneal colicky pain with suspected or confirmed nephrolithiasis during the main treatment period were assessed.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 1 | 0 | 0

29. Secondary Outcome: Number of Patients Treated With 30 mg/Day or 45 mg/Day IMU-838 as Compared to Placebo Who Experienced at Least One of the Following AEs:
Description: * Neutropenia
  * Lymphopenia
  * Diarrhea
  * Alopecia
  * Hemorrhage
  * Abnormalities in alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), and total bilirubin with both elevations ˃1.5 x ULN and ≥35% elevated compared to Baseline
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants
  Neutropenia | 0 | 0 | 1
  Lymphopenia | 0 | 0 | 0
  Diarrhea | 0 | 0 | 0
  Alopecia | 3 | 1 | 0
  Hemorrhage | 0 | 0 | 0
  ALT >1.5 x ULN AND representing a % change from Baseline ≥35% | 2 | 4 | 5
  AST >1.5 x ULN AND representing a % change from Baseline ≥35% | 1 | 3 | 4
  GGT >1.5 x ULN AND representing a % change from Baseline ≥35% | 3 | 2 | 1
  Total bilirubin >1.5 x ULN AND representing a % change from Baseline ≥35% | 0 | 0 | 0

30. Secondary Outcome: 12-lead Electrocardiogram (ECG): Heart Rate
Description: The 12-lead ECG was recorded in supine position after at least 5 minutes at rest using the local standard ECG machine. The ECG was analyzed qualitatively (normal or abnormal, if abnormal clinically significant [yes/no]). The heart rate, PQ-, QRS-, and QT intervals, as well as the heart rate-corrected QTc interval (according to Bazett's formula) were determined. All procedures were done according to local practice.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Median (Full Range); unit: beats per minute
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
beats per minute
  Screening 1 | 67.0 [45 to 100] | 68.0 [51 to 93] | 67.0 [46 to 97]
  Week 24: number analyzed (Participants) | 66 | 64 | 64
  Week 24 | 69.5 [46 to 120] | 69.0 [43 to 116] | 70.0 [46 to 105]

31. Secondary Outcome: 12-lead Electrocardiogram (ECG): PQ-interval
Description: as for outcome 30
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Median (Full Range); unit: msec
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
msec
  Screening 1 | 147.0 [95 to 448] | 140.0 [87 to 200] | 150.0 [95 to 200]
  Week 24: number analyzed (Participants) | 66 | 64 | 64
  Week 24 | 146.5 [77 to 247] | 146.0 [100 to 213] | 150.5 [92 to 202]

32. Secondary Outcome: 12-lead Electrocardiogram (ECG): QRS-interval
Description: as for outcome 30
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Median (Full Range); unit: msec
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
msec
  Screening 1 | 90.0 [60 to 148] | 86.0 [60 to 135] | 90.0 [66 to 112]
  Week 24: number analyzed (Participants) | 66 | 64 | 64
  Week 24 | 90.0 [60 to 128] | 86.0 [60 to 120] | 91.0 [60 to 113]

33. Secondary Outcome: 12-lead Electrocardiogram (ECG): QT-interval
Description: as for outcome 30
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Median (Full Range); unit: msec
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
msec
  Screening 1 | 383.0 [310 to 514] | 380.0 [320 to 447] | 387.0 [335 to 448]
  Week 24: number analyzed (Participants) | 66 | 64 | 64
  Week 24 | 376.5 [71 to 472] | 374.5 [286 to 472] | 385.0 [310 to 448]

34. Secondary Outcome: 12-lead Electrocardiogram (ECG): Heart Rate-corrected QTc Interval (According to Bazett's Formula)
Description: as for outcome 30
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Median (Full Range); unit: msec
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
msec
  Screening 1 | 407.0 [325 to 500] | 404.0 [340 to 483] | 410.0 [361 to 468]
  Week 24: number analyzed (Participants) | 66 | 64 | 64
  Week 24 | 407.0 [77 to 478] | 404.0 [283 to 467] | 409.0 [353 to 483]

35. Secondary Outcome: Physical Examination
Description: Physical examinations covered the following body systems: general appearance, skin, neck (including thyroid), throat, lungs, heart, abdomen, back, lymph nodes, extremities, vascular, neurological systems, and, if applicable, others. Any new clinically significant finding compared to Screening Visit 1 had to be documented as AE. Any clinically significant finding at Screening Visit 1 had to be documented in the medical history section of the eCRF.
  Patients with clinically significant findings in the physical examination post Day 0 are reported.
Time Frame: Up to 24 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 0 | 1 | 3

36. Secondary Outcome: Vital Signs: Height
Description: Height in centimeters was recorded without shoes. Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: at Screening
Population: Full analysis set
Measure: Median (Full Range); unit: cm
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
cm | 170.0 [154 to 198] | 167.0 [154 to 188] | 168.0 [149 to 192]

37. Secondary Outcome: Vital Signs: Weight (Absolute Change From Baseline at Week 24)
Description: Weight in kilograms was recorded without shoes. Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: Baseline and 24 weeks
Population: Patients with observations.
Measure: Median (Full Range); unit: kg
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 66 | 65 | 64
kg | 0.00 [-18.2 to 8.6] | 0.00 [-7.0 to 7.5] | 0.00 [-11.0 to 12.5]

38. Secondary Outcome: Vital Signs: Body Temperature (ºC) (Absolute Change From Baseline at Week 24)
Description: Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: Baseline and 24 weeks
Population: Patients with observations.
Measure: Median (Full Range); unit: °C
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 67 | 65 | 64
°C | 0.00 [-0.8 to 1.6] | 0.00 [-0.7 to 0.7] | 0.00 [-0.8 to 0.4]

39. Secondary Outcome: Vital Signs: Respiratory Rate (Absolute Change From Baseline at Week 24)
Description: Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: Baseline and 24 weeks
Population: Patients with observations
Measure: Median (Full Range); unit: breaths/min
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 67 | 65 | 64
breaths/min | 0.0 [-4 to 6] | 0.0 [-6 to 4] | 0.0 [-3 to 9]

40. Secondary Outcome: Vital Signs: Pulse Rates (Absolute Change From Baseline at Week 24)
Description: Pulse had to be measured with the patient in a seated position, after at least 5 minutes at rest.
  Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: Baseline and 24 weeks
Population: Patients with observations
Measure: Median (Full Range); unit: beats per minute
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 67 | 65 | 64
beats per minute | 0.0 [-24 to 16] | 0.0 [-30 to 24] | -1.0 [-18 to 22]

41. Secondary Outcome: Vital Signs: Systolic and Diastolic Blood Pressures (Absolute Change From Baseline at Week 24)
Description: Blood pressure (systolic and diastolic) had to be measured with the patient in a seated position, after at least 5 minutes at rest.
  Changes in vital signs judged by the investigator as clinically significant were to be reported as an AE.
Time Frame: Baseline and 24 weeks
Population: Patients with observations
Measure: Median (Full Range); unit: mmHg
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 67 | 65 | 64
mmHg
  Systolic blood pressure | 0.0 [-36 to 20] | 0.0 [-30 to 30] | 0.0 [-22 to 30]
  Diastolic blood pressure | 0.0 [-25 to 22] | 0.0 [-20 to 30] | 0.0 [-26 to 20]

42. Secondary Outcome: Micro Ribonucleic Acid (miR)-122 Expression
Description: The fold change in miR-122 from pre dose to 4 hours post dose was assessed.
Time Frame: Change from Baseline to 4 hours after first dose
Population: Patients with observations.
Measure: Median (Full Range); unit: fold change
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 67 | 67
fold change | 0.727 [0.12 to 63.23] | 0.991 [0.19 to 53.75] | 0.946 [0.12 to 50.11]

43. Secondary Outcome: Presence of John Cunningham Virus (JCV) Deoxyribonucleic Acid (DNA) in Urine in Patients With Detectable JCV-DNA in Urine
Description: The presence of JCV-DNA in urine in patients with detectable JCV-DNA in urine at Screening Visit 1, at Week 24, and at end-of-study (EoS) was determined.
Time Frame: At Screening Visit 1, at Week 24, and at EoS visit (EoS visit 30 days (+14 days) after last IMP intake)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants
  Screening 1: number analyzed (Participants) | 69 | 68 | 67
  Screening 1 | 32 | 27 | 29
  Week 24: number analyzed (Participants) | 65 | 62 | 63
  Week 24 | 27 | 16 | 18
  End-of-study: number analyzed (Participants) | 1 | 3 | 4
  End-of-study | 0 | 1 | 1

44. Secondary Outcome: Time to Treatment Discontinuation for Any Reason
Description: The time to treatment discontinuation up to Week 24 for any reason was determined.
Time Frame: Up to 24 weeks
Population: Patients with observations
Measure: Median (Full Range); unit: days
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 2 | 4 | 5
days | 106.5 [43 to 170] | 66.5 [47 to 178] | 98.0 [85 to 139]

45. Secondary Outcome: Rate of Treatment Discontinuations up to Week 24
Description: The discontinuation rate during the main treatment period was assessed.
Time Frame: at Week 24
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Participants | 2 | 4 | 5

46. Secondary Outcome: Population Pharmacokinetics: Minimum IMU-838 Plasma Concentration Over the Dosing Interval (Cmin)
Description: One single measurement between 3 and 10 hours post-dose. Population pharmacokinetics have not been reported yet.
Time Frame: At Week 6 (3-10 hours post-dose)
Population: Data have not yet been analyzed.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

47. Secondary Outcome: Population Pharmacokinetics: Maximum IMU-838 Plasma Concentration Over the Dosing Interval (Cmax)
Description: One single measurement between 3 and 10 hours post-dose. Population pharmacokinetics have not been reported yet.
Time Frame: At Week 6 (3-10 hours post-dose)
Population: Data have not yet been analyzed.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

48. Secondary Outcome: Population Pharmacokinetics: Area Under the IMU-838 Plasma Concentration-time Curve Over the Dosing Interval (AUC0-τ)
Description: One single measurement between 3 and 10 hours post-dose. Population pharmacokinetics have not been reported yet.
Time Frame: At Week 6 (3-10 hours post-dose)
Population: Data have not yet been analyzed.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

49. Secondary Outcome: Population Pharmacokinetics: IMU-838 Apparent Clearance Following Oral Dosing (CL/F)
Description: One single measurement between 3 and 10 hours post-dose. Population pharmacokinetics have not been reported yet.
Time Frame: At Week 6 (3-10 hours post-dose)
Population: Data have not yet been analyzed.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

50. Secondary Outcome: Population Pharmacokinetics: IMU-838 Apparent Volume of Distribution (V/F)
Description: One single measurement between 3 and 10 hours post-dose. Population pharmacokinetics have not been reported yet.
Time Frame: At Week 6 (3-10 hours post-dose)
Population: Data have not yet been analyzed.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

51. Secondary Outcome: Plasma Trough Levels of IMU-838
Description: Plasma trough levels of IMU-838 were assessed at Day 7 and at Weeks 6, 12, 18, and 24.
Time Frame: At Day 7 and Weeks 6, 12, 18, and 24
Population: Safety set
Measure: Median (Full Range); unit: μg/mL
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day)
Number analyzed (Participants) | 71 | 69
μg/mL
  Day 7: number analyzed (Participants) | 70 | 69
  Day 7 | 2.155 [0.90 to 8.96] | 3.100 [0.12 to 7.89]
  Week 6: number analyzed (Participants) | 71 | 66
  Week 6 | 4.320 [0.00 to 15.70] | 6.240 [0.00 to 18.30]
  Week 12: number analyzed (Participants) | 69 | 67
  Week 12 | 4.160 [0.00 to 12.40] | 5.420 [0.00 to 14.00]
  Week 18: number analyzed (Participants) | 70 | 65
  Week 18 | 4.165 [0.00 to 12.10] | 5.990 [0.00 to 15.00]
  Week 24: number analyzed (Participants) | 67 | 64
  Week 24 | 4.010 [0.00 to 8.14] | 5.700 [0.00 to 16.30]

52. Secondary Outcome: Changes From Baseline in Th1 Lymphocyte Subset as Measured by Flow Cytometry
Description: Changes from Baseline in lymphocyte subsets were listed only; no descriptive statistics by treatment arm were calculated.
Time Frame: At Weeks 6 and 24 (in selected Biomarker Centers only)
Population: Changes from Baseline in Th1 lymphocyte subsets were listed only; no descriptive statistics by treatment arm were calculated.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

53. Secondary Outcome: Changes From Baseline in Th17 Lymphocyte Subset as Measured by Flow Cytometry
Description: as for outcome 52
Time Frame: At Weeks 6 and 24 (in selected Biomarker Centers only)
Population: Changes from Baseline in Th17 lymphocyte subsets were listed only; no descriptive statistics by treatment arm were calculated.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

54. Secondary Outcome: Changes From Baseline in Treg Lymphocyte Subset as Measured by Flow Cytometry
Description: as for outcome 52
Time Frame: At Weeks 6 and 24 (in selected Biomarker Centers only)
Population: Changes from Baseline in Treg lymphocyte subsets were listed only; no descriptive statistics by treatment arm were calculated.
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

55. Secondary Outcome: Changes From Baseline in Serum Neurofilament
Description: The percentage change from Baseline in serum neurofilament was calculated.
Time Frame: At Week 6 and Week 24
Population: Safety data set
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
percent change
  Week 6 | -4.0 [-10.0 to 8.0] | -1.0 [-12.0 to 8.0] | 8.0 [-5.0 to 15.0]
  Week 24: number analyzed (Participants) | 67 | 64 | 64
  Week 24 | -17.0 [-24.0 to -7.0] | -20.5 [-29.0 to -13.0] | 6.5 [-11.0 to 25.0]

56. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: The TSQM is a reliable and valid instrument to assess patients' satisfaction with medication comprising 14 items across 4 domains: side effects, performance, convenience and global satisfaction. All items have 5 to 7 possible answers, except for item 4 (2 answers).
  Item scores for each domain are summed and transformed to a scale from 0 (extremely dissatisfied) to 100 (extremely satisfied).
Time Frame: assessed at 6 weeks, 24 weeks, and end of study visit (EoS visit 30 days [+14 days] after last IMP intake), reported at Week 6 and Week 24
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: score
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
score
  Effectiveness at Week 6 | 62.45 (16.73) | 67.16 (15.44) | 60.55 (15.66)
  Effectiveness at Week 24: number analyzed (Participants) | 69 | 65 | 64
  Effectiveness at Week 24 | 66.43 (14.61) | 71.28 (17.58) | 61.72 (15.27)
  Side effects at Week 6 | 92.70 (16.53) | 96.02 (12.21) | 95.29 (13.65)
  Side effects at Week 24: number analyzed (Participants) | 69 | 65 | 64
  Side effects at Week 24 | 97.10 (9.37) | 97.41 (11.25) | 95.41 (12.99)
  Convenience at Week 6 | 82.62 (13.03) | 81.48 (15.40) | 80.59 (13.98)
  Convenience at Week 24: number analyzed (Participants) | 69 | 65 | 64
  Convenience at Week 24 | 82.12 (12.55) | 84.18 (14.66) | 79.69 (13.13)
  Global satisfaction at Week 6 | 67.30 (18.34) | 70.29 (15.34) | 63.87 (16.93)
  Global satisfaction at Week 24: number analyzed (Participants) | 69 | 65 | 64
  Global satisfaction at Week 24 | 70.07 (16.13) | 75.05 (17.87) | 66.29 (15.04)

57. Secondary Outcome: Difference Between 30 mg/Day IMU-838 and Placebo, 45 mg/Day IMU-838 and Placebo, and 30 mg/Day and 45 mg/Day IMU-838 for Brain Atrophy.
Description: This endpoint was added in statistical analysis plan Version 2.0. Results of the brain atrophy analysis included biologically implausible changes (including changes of more than 1% over 24 weeks) in all treatment groups. Hence, the brain volume changes were considered technically inadequate for any conclusions of a treatment effect of IMU-838 versus placebo.
Time Frame: Baseline, Week 6, Week 12, Week 18, and Week 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
Number analyzed (Participants) | 71 | 69 | 69
Percent change | NA (NA) — Results of the brain atrophy analysis included biologically implausible changes (including changes of more than 1% over 24 weeks) in all treatment groups. Hence, the brain volume changes were considered technically inadequate for any conclusions of a treatment effect of IMU-838 versus placebo. | NA (NA) — Results of the brain atrophy analysis included biologically implausible changes (including changes of more than 1% over 24 weeks) in all treatment groups. Hence, the brain volume changes were considered technically inadequate for any conclusions of a treatment effect of IMU-838 versus placebo. | NA (NA) — Results of the brain atrophy analysis included biologically implausible changes (including changes of more than 1% over 24 weeks) in all treatment groups. Hence, the brain volume changes were considered technically inadequate for any conclusions of a treatment effect of IMU-838 versus placebo.

ADVERSE EVENTS:
Time Frame: Main treatment period (24 weeks)
Arm/Group | IMU-838 (30 mg/Day) | IMU-838 (45 mg/Day) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/71 | 0/69 | 1/69
Other Adverse Events (participants affected / at risk) | 6/71 | 7/69 | 7/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMU-838 (30 mg/Day) (N=71) | IMU-838 (45 mg/Day) (N=69) | Placebo (N=69)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMU-838 (30 mg/Day) (N=71) | IMU-838 (45 mg/Day) (N=69) | Placebo (N=69)
Nasopharyngitis (Infections and infestations) | 3 (5) | 5 (7) | 3 (4)
Headache (Nervous system disorders) | 3 (3) | 4 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03846219/Prot_SAP_000.pdf